CLINICAL TRIAL: NCT01409525
Title: Observational, Prospective, Exploratory Study to Evaluate the Rate of Microbial Colonization Over Native Calcified Cardiac Valves
Brief Title: Rate of Microbial Colonization Over Native Calcified Cardiac Valves
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Liran Shani, Rambam Health Care Campus- cardiac surgery department
Other Study IDs: RMB-0233.CTIL
Record Dates: First submitted 2011-07-28; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Degenerative Cardiac Valve Disease; Coronary Artery Bypass Surgery Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cardiac valve tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac surgery patients

SUMMARY:
The purpose of this observational, exploratory study in patients undergoing any cardiac valve replacement or repair is to assess the rate of bacterial colonization over native degenerative calcified cardiac valves.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the subject or his/her legal guardian before any assessment is performed
* Male or Female subject, 50 years or older
* Subjects are scheduled to go through any cardiac valve replacement or repair due to degenerative calcified process. For control, subjects with no evidence of valve disease

Exclusion Criteria:

* Subjects have an established or indicated history of IE.
* Subjects have complaint that might indicate IE- intermittent fever and physical finding according to IE diagnosis criteria (not including a heart murmur)
* Subjects are current users or have a close history of drug abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 200 eligible adult subjects, scheduled to undergo elective cardiac surgery in RAMBAM medical center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
To asses the rate of bacterial colonization over degenerative cardiac valves and to discover whether there is a link to a specific micro-organism. | Patients will be followed for the duration of their hospitalization, average of 5 days.

SECONDARY OUTCOMES:
Correlation between baseline demographic, clinical and laboratory parameters to degenerative cardiac valve disease | Patients will be followed for the duration of their hospitalization, average of 5 days.
  Baseline demographic, clinical and laboratory parameters such as age, gender, medical history, complete blood count and biochemistry profile will be compared between research group (degenerative cardiac valve disease) and control group (Isolated coronary artery bypass graft surgery patients) by means of multivariate analysis and pattern recognition techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Liran Shani, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel